CLINICAL TRIAL: NCT06826534
Title: At-Home Cardiac Rehabilitation for Adolescents at Risk for Heart Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Jennifer Su, Assistant Professor, Keck School of Medicine, University of Southern California, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHLA-22-00323
Record Dates: First submitted 2025-01-31; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Cardiovascular Complication; Chemotherapeutic Toxicity
Keywords: anthracycline exposure; cancer survivors; physical activity; pediatric oncology; cardiac rehabilitation
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental)
  Interventions: Behavioral: Cardio-oncology rehabilitation

INTERVENTIONS:
Behavioral: Cardio-oncology rehabilitation — Least 60 minutes of physical activity each day including vigorous-intensity and strengthening activities at least 3 days per week

SUMMARY:
The goal of this clinical trial is to explore the impact that an at-home cardio-oncology rehabilitation (CORE) may have on short-term cardiovascular fitness and psychosocial wellness in pediatric cancer survivors. The main question it aims to answer are

* To evaluate the efficacy of an at-home CORE model on short-term cardiovascular fitness and psychosocial wellbeing in adolescent cancer survivors.
* To evaluate the exercise adherence rate among adolescents at risk for heart failure and assess barriers to compliance.
* To explore which specific CORE resources are of most value to patients in creating sustainable healthy lifestyle modifications.
* Hypothesis: Pediatric cancer survivors who implement exercise and dietary recommendations will demonstrate improvement in cardiovascular fitness and general wellness. A multidisciplinary team approach can facilitate adherence to a moderately rigorous exercise prescription, and thus enhance the health benefits of a CORE program at CHLA.

Participants will undergo cardiovascular studies and a quality-of-life survey prior to exercise intervention, and at the end of the 6-month study period.

ELIGIBILITY:
INCLUSION CRITERIA

* Patients aged of 10-21 years at enrollment
* Parent/legal guardian available for consent (if applicable), and patient available for assent and consent
* History of anthracycline exposure +/- radiation
* Currently in remission, with at least 6 months off chemotherapy
* Able to perform CPET
* Baseline CPET with VO2 <80% (at start of study, or CPET at CHLA after January 2020)
* Smartphone compatible with Fitbit (own or parent/legal guardian's)
* Ability to complete and send diary and Fitbit information on a weekly basis
* Ability to participate in monthly virtual check-in visits
* Baseline activity prior to intervention <30min/day, 2x/week

EXCLUSION CRITERIA

* Inability to obtain consent/assent
* Unable to accurately perform quality of life survey independently
* No other primary medical diagnosis (e.g., Down Syndrome, Wolff-Parkinson-White Syndrome, congenital heart disease) or history of cardiothoracic surgery
* Contraindication to moderate activity (>3 METs). Examples include history of malignant arrhythmias, exercise-induced syncope, severe symptoms of HF (NYHA IV, ACC/AHA Stage D)
* Unable to perform CPET, echocardiogram, EKG, or obtain laboratory studies
* Unable to perform mild activity for at least 0.5h/day and at least 2x/week
* Unable to come to hospital for study visits at 0 and 6 months
* Unable to complete study-related surveys
* Unable to complete and send diary and Fitbit information on a weekly basis
* Unable to check-in monthly on virtual platform
* On beta blockade
* Pregnancy

Ages: 0 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in cardiovascular fitness after completion of a 6-month exercise intervention. | Baseline to 6 months
  Peak VO2% (exercise capacity) as measured by cardiopulmonary exercise testing.
Change in cardiovascular fitness after completion of a 6-month exercise intervention. | Baseline to 6 months
  Ve/VCO2 slope (predictor of cardiac mortality) as measured by cardiopulmonary exercise testing.
Change in cardiovascular fitness after completion of a 6-month exercise intervention. | Baseline to 6 months
  Chronotropic response (heart rate response to exercise) as measured by cardiopulmonary exercise testing.
Change in cardiovascular fitness after completion of a 6-month exercise intervention. | Baseline to 6 months
  Blood pressure response to exercise as measured by cardiopulmonary exercise testing.
Change in cardiac function after completion of a 6-month exercise intervention. | Baseline to 6 months
  Cardiac function will be assessed via echocardiogram.
Change in cardiac rhythm after completion of a 6-month exercise intervention. | Baseline to 6 months
  Cardiac rhythm will be assessed via EKG.
Change in cardiac stress after completion of a 6-month exercise intervention. | Baseline to 6 months
  Cardiac stress will be assessed via NT-proBNP level.
Average change in triglyceride level as measured from baseline to 6 months. | Baseline to 6 months
  Triglyceride (mg/dL) will be measured.
Average change in total cholesterol level as measured from baseline to 6 months. | Baseline to 6 months
  Total cholesterol (mg/dL) will be measured.
Average change in high density lipoprotein level as measured from baseline to 6 months. | Baseline to 6 months
  High density lipoprotein (HDL) (mg/dL) will be measured.
Average change in low density lipoprotein as measured from baseline to 6 months. | Baseline to 6 months
  Low density lipoprotein (LDL) (mg/dL) will be measured.
Average change in very low density lipoprotein as measured from baseline to 6 months. | Baseline to 6 months
  Very low density lipoprotein (VLDL) (mg/dL) will be measured.

SECONDARY OUTCOMES:
Average change in reported quality of life from baseline to 6 months | Baseline to 6 months
  PedsQL(TM) Measurement Model will be used, which assesses physical, emotional, social, school functioning domains.
Percent of participants with improvement in healthy lifestyle habits from baseline to 6 months | Baseline to 6 months
  Lifestyle habits will be assessed via exercise and dietary surveys completed by each participant.
Average change in activity level from baseline to 6 months | Baseline to 6 months
  Activity levels will be assessed via exercise surveys as well as continuous FitBit(TM) activity data which will include weekly number of steps, average calorie burn, days of exercise, minute in activity, and average sleep time.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Su, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No